CLINICAL TRIAL: NCT02628327
Title: Factors Influencing Patient Satisfaction in a Glaucoma Population
Acronym: FIPSS
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Jonathon Myers, Principle Investigator, Wills Eye
Other Study IDs: 15-496E
Record Dates: First submitted 2015-08-06; First posted 2015-12-11 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: glaucoma care; quality of life; patient satisfaction
MeSH Terms: conditions — Glaucoma; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma subjects: Survey given to all glaucoma subjects agreening to study.

SUMMARY:
1. To administer a questionnaire to patients seen by Wills Eye Glaucoma Department physicians at Wills Eye Hospital assessing satisfaction with their office visit, vision related quality of life, and related issues.
2. To collect and de-identify information from each participant's medical chart related to their care including information pertaining to demographics, disease severity, and prior and current treatment
3. To assess the correlations between demographic factors, vision related quality of life, eye disease, and treatments with patient satisfaction survey responses.

DETAILED DESCRIPTION:
This prospective study aims to recruit up to 250 patients being seen by glaucoma specialists at Wills Eye Hospital. Informed consent will be obtained prior to the office visit. Patients will complete a satisfaction survey with a few additional questions about themselves and their vision. Electronic health records (EHR) will be used to collect race, gender, age, glaucoma diagnosis, current and prior treatments, timing of appointment and care, visual acuity and field data, and distance to patient's home. Additional information captured will include weather, time of day, day of week.

In addition to completing the questionnaire subjects will be asked to provide their name and date of birth. Trained research staff members will use this information to find patients on the EHR system. A research assistant will later abstract information from the patient's EHR. This information will be tagged to the survey by a unique identifier, but all patient identity related information will be removed, including name and date of birth. Patients will be made aware that research staff will be retrieving their protected health information (PHI) for the purpose of this study through the consent form.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years; patients who have a scheduled appointment at with a glaucoma specialist at Wills Eye Hospital; diagnosis of glaucoma or glaucoma suspect

Exclusion Criteria:

Children under the age of 18; inability to give informed consent; patients who are physically and/or mentally incapable of filling out a paper survey; patients who are not literate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma or glaucoma suspect
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life assessment | 6 months
  Correlate demographic factors to vision related quality of life, eye disease and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Myers, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript has been submitted to the Journal of Medical Quality